CLINICAL TRIAL: NCT01402895
Title: The Effect Of A Neurodynamic Treatment On Nerve Conduction In Clients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-541
Record Dates: First submitted 2011-07-22; First posted 2011-07-26 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2011-07

CONDITIONS: Low Back Pain
Keywords: Nerve conduction; H-reflex, mobilizations; with neurodynamic component
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobilizations (Active Comparator): The physiotherapist will perform mobilizations to the L-spine and SI joints with the participant in a specific position.
  Interventions: Other: Mobilizations
- Exercise (Active Comparator): The physiotherapist will teach the participant how to tighten the transversus abdominus muscle. The participant will be asked to do a series of these exercises.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Transversus abdominus exercise
  Arms: Exercise
Other: Mobilizations — The physiotherapist will perform mobilizations to the L-spine and SI joints with the participant in a specific position.
  Arms: Mobilizations

SUMMARY:
The purpose of this study is to determine if a certain treatment for low back pain can change the way nerves in the leg send messages. Specifically, the investigators will examine whether a particular type of physical therapy treatment for individuals with low back pain (neurodynamic techniques) changes the speed that nerves send/receive signals to/from the leg, as compared to a different physical therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years and older
* Participants who can speak English and read, understand, and fill out the consent form and questionnaires
* Participants will have a certain level of low back pain graded numerically, with or without radiation to the leg
* Clinical decision (by same individual) as safe to participate in study based on subjective history and objective examination.

Exclusion Criteria:

* An inability to tolerate sitting for 10 minutes
* Nerve conduction disorders diagnosed by a physician such as, diabetes or MS
* Current participant in an investigational drug study (within past 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in nerve conduction studies | Change from baseline after intervention, on average 1.5 hours after baseline measure
  Motor conduction of the tibial nerve; Sensory conduction of the sural nerve; H-reflex, H:M ratio (soleus muscle)

SECONDARY OUTCOMES:
Change of knee extension in sitting slump test | Change from baseline after intervention, on average 1.5 hours after baseline measure
Change in score of Visual Analog Scale for pain | Change from baseline after intervention, on average 1.5 hours after baseline measure

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Galea, PhD, Study Director — McMaster University; Joy MacDermid, PhD, Study Chair — McMaster University; Linda Woodhouse, PhD, Study Chair — University of Alberta; Anita Gross, MSc, Study Chair — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Breig A, Troup JD. Biomechanical considerations in the straight-leg-raising test. Cadaveric and clinical studies of the effects of medial hip rotation. Spine (Phila Pa 1976). 1979 May-Jun;4(3):242-50. doi: 10.1097/00007632-197905000-00011. PMID 157532
- [Background] Butler, D.S. (1991). SLR, The Slump Test in Mobilisation of the Nervous System (pp.130-135, 139-146). London (UK): Elsevier Limited.
- [Background] Cyriax J. Perineuritis. Br Med J. 1942 May 9;1(4244):578-80. doi: 10.1136/bmj.1.4244.578. No abstract available. PMID 20784219
- [Background] DeLeo JA. Basic science of pain. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:58-62. doi: 10.2106/JBJS.E.01286. PMID 16595445
- [Background] Gelberman RH, Szabo RM, Williamson RV, Hargens AR, Yaru NC, Minteer-Convery MA. Tissue pressure threshold for peripheral nerve viability. Clin Orthop Relat Res. 1983 Sep;(178):285-91. PMID 6883862
- [Background] Kimura, J. (1983). Tibial nerve, Sural nerve, The H-reflex and other late responses., Electrodiagnosis in Diseases of Nerve and Muscle: Principles and Practice. (pp. 125-127, 130-134, 379-385). U.S.A.: F. A. Davis Company.
- [Background] Lundborg G, Rydevik B. Effects of stretching the tibial nerve of the rabbit. A preliminary study of the intraneural circulation and the barrier function of the perineurium. J Bone Joint Surg Br. 1973 May;55(2):390-401. No abstract available. PMID 4707307
- [Background] Mahmud MA, Merlo AR, Gomes I, Becker J, Nora DB. [Relationship between adverse neural tension and nerve conduction studies in patients with symptoms of the carpal tunnel syndrome]. Arq Neuropsiquiatr. 2006 Jun;64(2A):277-82. doi: 10.1590/s0004-282x2006000200019. Epub 2006 Jun 9. Portuguese. PMID 16791369
- [Background] Maitland GD. Negative disc exploration: positive canal signs. Aust J Physiother. 1979 Jul;25(3):129-34. doi: 10.1016/S0004-9514(14)61220-4. PMID 25026403
- [Background] Nakamichi K, Tachibana S. Restricted motion of the median nerve in carpal tunnel syndrome. J Hand Surg Br. 1995 Aug;20(4):460-4. doi: 10.1016/s0266-7681(05)80153-6. PMID 7594983
- [Background] Ogata K, Naito M. Blood flow of peripheral nerve effects of dissection, stretching and compression. J Hand Surg Br. 1986 Feb;11(1):10-4. doi: 10.1016/0266-7681(86)90003-3. PMID 3958526
- [Background] Schaafsma L, Sun H, Zochodne D. Exogenous opioids influence the microcirculation of injured peripheral nerves. Am J Physiol. 1997 Jan;272(1 Pt 2):H76-82. doi: 10.1152/ajpheart.1997.272.1.H76. PMID 9038924
- [Background] Shacklock, M. (1995). Neurodynamics. Physiotherapy, 81, 9-16.
- [Background] Shacklock, M. (2005a). Clinical neurodynamics: A new system of musculoskeletal treatment (pp. 2-29, 98-104, 154-158). London (UK): Elsevier Butterworth Heinemann.
- [Background] Shacklock M. Improving application of neurodynamic (neural tension) testing and treatments: a message to researchers and clinicians. Man Ther. 2005 Aug;10(3):175-9. doi: 10.1016/j.math.2005.03.001. Epub 2005 Apr 20. No abstract available. PMID 16038853
- [Background] Spadoni GF, Stratford PW, Solomon PE, Wishart LR. The evaluation of change in pain intensity: a comparison of the P4 and single-item numeric pain rating scales. J Orthop Sports Phys Ther. 2004 Apr;34(4):187-93. doi: 10.2519/jospt.2004.34.4.187. PMID 15128188
- [Background] Stretanski MF. H-reflex latency and nerve root tension sign correlation in fluoroscopically guided, contrast-confirmed, translaminar lumbar epidural steroid-bupivacaine injections. Arch Phys Med Rehabil. 2004 Sep;85(9):1479-82. doi: 10.1016/j.apmr.2003.09.024. PMID 15375820
- [Background] WOODHALL B, HAYES GJ. The well-legraising test of Fajersztajn in the diagnosis of ruptured lumbar intervertebral disc. J Bone Joint Surg Am. 1950 Oct;32 A(4):786-92. No abstract available. PMID 14784487
- [Background] Zochodne DW, Ho LT. Stimulation-induced peripheral nerve hyperemia: mediation by fibers innervating vasa nervorum? Brain Res. 1991 Apr 12;546(1):113-8. doi: 10.1016/0006-8993(91)91165-w. PMID 1855142
- [Background] Zochodne DW, Huang ZX, Ward KK, Low PA. Guanethidine-induced adrenergic sympathectomy augments endoneurial perfusion and lowers endoneurial microvascular resistance. Brain Res. 1990 Jun 11;519(1-2):112-7. doi: 10.1016/0006-8993(90)90067-l. PMID 2397398
- [Background] Zochodne DW, Low PA. Adrenergic control of nerve blood flow. Exp Neurol. 1990 Sep;109(3):300-7. doi: 10.1016/s0014-4886(05)80021-4. PMID 2285433